CLINICAL TRIAL: NCT01298830
Title: GLP-1 CellBeads® for the Treatment of Stroke Patients With Space-occupying Intracerebral Hemorrhage
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Need for improvement of study medication. Safety data collected sufficient. No further gain in knowledge expected.
Sponsor: CellMed AG, a subsidiary of BTG plc. (Industry)
Responsible Party: Dr. med. Peter Geigle / CEO, CellMed AG
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CM GLP-1/01; 2007-004516-31 (EudraCT Number)
Record Dates: First submitted 2011-02-15; First posted 2011-02-18 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2013-03

CONDITIONS: Intracerebral Hemorrhage (ICH)
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GLP-1 CellBeads (Experimental)
  Interventions: Drug: GLP-1 CellBeads

INTERVENTIONS:
Drug: GLP-1 CellBeads — GLP-1 CellBeads are alginate microcapsules containing allogenic mesenchymal cells, transfected to secrete Glucagon like peptide-1. By implantation into brain tissue cavity after surgical evacuation of the hematoma, a volume of 500μl GLP-1 CellBeads which equals approximately 2330 GLP-1 CellBeads resulting in a total number of approximately 7.8 million cells is administered to the patient. The cells are removed by second surgery after a 14 days treatment period.

SUMMARY:
The objective of this study is to assess the safety of GLP-1 CellBeads® in patients with space-occupying intracerebral hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of intracerebral hemorrhage or subarachnoid hemorrhage in conjunction with ICH by cranial computed tomography (CCT) or Magnetic Resonance Tomography (MRT)
* Patients who need by judgement of a clinical neurologist or neurosurgeon surgical removal of the blood clot due to its space-occupying effects
* Age greater or equal 18 years for men
* Age greater or equal 18 years for women if confirmed infertility (e.g. hysterectomy or surgical sterilisation at least 3 months before study start)
* For all other women age greater or equal 50 years with last menstrual bleeding at least one year before study start
* Minimum hematoma diameter of 2 cm as measured in baseline CCT or MRT
* Signed, written informed consent of patient or consent/assertion from the patient's legally acceptable representative/affiliated if the patient is unable to provide informed consent

Exclusion Criteria:

* Participation in any other clinical trial within the past 3 months or ongoing
* Occurrence of inconsistency with initial diagnosis at baseline during surgery of the patient leading to unfulfilled inclusion criterion Hemorrhage secondary to tumour or trauma
* Patients with a cerebellar hemorrhage or extension of a supratentorial hemorrhage into the brainstem
* Patients with severe pre-existing physical or mental disability or severe comorbidity that interferes with the assessment of outcome
* Allergy to contrast media (MRT)
* Acute infection
* Muscular, neurological, or vascular insufficiency of the respective tissue
* Polypropylene incompatibility
* Acute immunosuppressive medication
* Patient after organ transplantation
* Patient with immune depression
* Patients with a high probability of spontaneous recovery or showing rapidly improving signs
* Patients with extensive intracranial hemorrhages or with deep hemispheric localisation of the clots
* Patients whose diagnosis of ICH is uncertain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The objective of this study is to assess the safety of GLP-1 CellBeads® in patients with space-occupying intracerebral hemorrhage | 6 months

SECONDARY OUTCOMES:
Neurological conditions | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Brinker, Prof. Dr.med., Study Chair — International Neuroscience Institute Hanover
Locations (6):
- Germany (6):
  - Neurochirurgische Klinik und Neurologische Klinik des Universitätsklinikums Heidelberg, Heidelberg, Baden-Wurttemberg
  - Neurochirurgische Klinik der Universität Erlangen-Nürnberg, Erlangen, Bavaria
  - Klinik für Neurochirurgie Klinikum Bogenhausen Akademisches Lehrkrankenhaus der Technischen Universität München, München, Bavaria
  - Klinikum Region Hannover Krankenhaus Nordstadt, Klinik für Neurologie, Hanover, Lower Saxony
  - International Neuroscience Institute, Hanover, Lower Saxony
  - Klinik für Neurochirurgie Medizinische Hochschule Hannover, Hanover, Lower Saxony